CLINICAL TRIAL: NCT06513559
Title: Anatomic Versus Reverse Shoulder Arthroplasty for Primary Glenohumeral Osteoarthritis: a Randomized Prospective Study
Brief Title: Anatomic Versus Reverse Shoulder Arthroplasty for Primary Glenohumeral Osteoarthritis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There was difficulty getting the study up and running with the site, staffing issues, completing a DTA and concern over sufficient patient population. The study was stopped without any enrollment. No results were obtained.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Joyce, Principle Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 159808
Record Dates: First submitted 2024-07-08; First posted 2024-07-22 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Glenohumeral Osteoarthritis
Keywords: glenohumeral osteoarthritis; reverse total shoulder arthroplasty; anatomic replacement; reverse replacement; range of motion; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Anatomic total shoulder replacement (Experimental): Anatomic replacement replaces the humeral head with a metal ball and the glenoid socket with a polyethylene glenoid component.
  Interventions: Device: Anatomic total shoulder replacement
- Reverse total shoulder replacement (Experimental): Reverse shoulder replacement reverses these implants with the polyethylene socket on the humeral side and the glenosphere going on the glenoid side.
  Interventions: Device: Reverse total shoulder replacement

INTERVENTIONS:
Device: Anatomic total shoulder replacement — Humeral head with a metal ball and the glenoid socket with a polyethylene glenoid component.
  Other Names: Arthrex Eclipse stem with a polyethylene glenoid.; Stryker perform stem with cortiloc glenoid; Enovis CS Edge stem with altivate anatomic glenoid; Exactech Equinoxe stem with cage anatomic glenoid
  Arms: Anatomic total shoulder replacement
Device: Reverse total shoulder replacement — Polyethylene socket on the humeral side and the glenosphere going on the glenoid side.
  Other Names: Arthrex Universe Reverse.; Stryker perform reverse; Enovis Altivate reverse; Exactech Equinoxe reverse
  Arms: Reverse total shoulder replacement

SUMMARY:
The primary goal of the investigators prospective randomized study is to determine whether reverse total shoulder arthroplasty (RTSA) have at least as good results as anatomic TSA (non-inferiority), in patients with glenohumeral osteoarthritis, without rotator cuff tears nor significant glenoid retroversion.

The secondary goals are 1) to evaluate whether RTSA eventually grants superior postoperative clinical and radiographic outcomes than anatomic TSA (superiority), 2) to determine whether RTSA is associated with fewer postoperative complications than anatomic TSA.

The devices being used in the research are an Arthrex Universe system (Arthrex Univers Reverse vs Arthrex Apex humeral stem or Eclipse stem with a polyethylene glenoid). They are FDA approved, commonly used, and used as indicated. The anatomic replacement replaces the humeral head with a metal ball and the glenoid socket with a polyethylene glenoid component. The reverse shoulder replacement reverses these implants with the polyethylene socket on the humeral side and the glenosphere going on the glenoid side.

In all cases, a deltopectoral incision will be used as the procedure type.

DETAILED DESCRIPTION:
Total anatomic shoulder arthroplasty (TSA) is an effective treatment of severe glenohumeral osteoarthritis, with significant improvement in shoulder pain and function. Concerns about glenoid loosening, associated with difficult revision procedures and disappointing outcomes, have however been raised.

Reverse total shoulder arthroplasty (RTSA) was designed to treat cuff tear arthropathy. Favorable early reports led to the expansion of using RTSA to treat other shoulder fractures as well as osteoarthritis with poor glenoid bone stock. Recent reports revealed excellent clinical results of RTSA for primary glenohumeral arthropathy with intact rotator cuff and a low rate of complications.

Retrospective studies comparing functional results - of anatomic TSA for treating glenohumeral osteoarthritis with RTSA for rotator cuff arthropathy - found equivalent or greater improvements in American Shoulder and Elbow Surgeons score (ASES) at >2-year follow-up. In a study comparing anatomic TSA to RTSA for the treatment of glenohumeral osteoarthritis with intact rotator cuffs, investigators have reported equivalent functional results at >2-year follow-up. However, this study could not eliminate biases, such that RTSA patients had higher preoperative glenoid retroversion than anatomic TSA patients.The investigators therefore hypothesize that, in patients treated for glenohumeral osteoarthritis, RTSA will render better functional outcomes than anatomic TSA, at 2 postoperative years. Many other studies have confirmed this hypothesis. Moreover, several studies revealed good long-term survivorship after RTSA.

There are no published prospective studies that compared 2-year functional outcomes of RTSA and anatomic TSA for the treatment of primary glenohumeral osteoarthritis with intact rotator cuffs and no excessive glenoid retroversion.

ELIGIBILITY:
Inclusion Criteria:

* Primary glenohumeral arthritis,
* Intact rotator cuff,
* No important glenoid bone loss (cf exclusion criteria),
* Patients between 60 and 85 years old (based on indications for RTSA)
* Informed Consent as documented by signature (Appendix Informed Consent Form).

Exclusion Criteria:

* B2 glenoid with > 80% posterior humeral head subluxation or greater 25 degrees neoglenoid retroversion,
* B3 and C type glenoids,
* Full thickness rotator cuff tear,
* Acute or malunited proximal humeral fracture,
* Chronic locked dislocation
* Rheumatoid arthritis,
* Revision surgery or surgical antecedents,
* Tumors,
* Axillary nerve damage,
* Non-functioning deltoid muscle,
* Glenoid vault deficiency precluding baseplate fixation,
* Infection and neuropathic joints,
* Known or suspected non-compliance, drug or alcohol abuse,
* Patients incapable of judgement or under tutelage,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, contraindication for CT scan etc. of the participant,

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons score | date of surgery
  Shoulder specific scoring system out of 100. A patient-reported score with visual analog scale for pain and functional subscales ranging from 0 (worse pain and function loss) to 50 (no pain and excellent function). Both scores are summed for a maximum score of 100.
American Shoulder and Elbow Surgeons score | 6 months after date of surgery
  Shoulder specific scoring system out of 100. A patient-reported score with visual analog scale for pain and functional subscales ranging from 0 (worse pain and function loss) to 50 (no pain and excellent function). Both scores are summed for a maximum score of 100.
American Shoulder and Elbow Surgeons score | 12 months after date of surgery
  Shoulder specific scoring system out of 100. A patient-reported score with visual analog scale for pain and functional subscales ranging from 0 (worse pain and function loss) to 50 (no pain and excellent function). Both scores are summed for a maximum score of 100.
American Shoulder and Elbow Surgeons score | 24 months after date of surgery
  Shoulder specific scoring system out of 100. A patient-reported score with visual analog scale for pain and functional subscales ranging from 0 (worse pain and function loss) to 50 (no pain and excellent function). Both scores are summed for a maximum score of 100.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Joyce, M.D., Principal Investigator — University of Utah Orthopaedics
Locations (1):
- University of Utah Orthopedics, Salt Lake City, Utah, United States